CLINICAL TRIAL: NCT03337165
Title: Safety/Efficacy of Intra-articular Administration of Autologous Tolerogenic Dendritic Cells for Treatment of Patients With Rheumatoid Arthritis
Brief Title: Autologous Tolerogenic Dendritic Cells for Treatment of Patients With Rheumatoid Arthritis
Acronym: TolDCfoRA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Russian Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Alexander A Ostanin, Head of Clinical Department, Russian Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IFCI-14/10/2016
Record Dates: First submitted 2017-11-03; First posted 2017-11-08 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Musculoskeletal Diseases; Joint Disease; Arthritis; Arthritis, Rheumatoid; Rheumatic Diseases; Connective Tissue Diseases; Autoimmune Diseases; Immune System Diseases
Keywords: Rheumatoid arthritis; Auto-immune disorders; Tolerogenic Dendritic Cells
MeSH Terms: conditions — Musculoskeletal Diseases; Joint Diseases; Arthritis; Arthritis, Rheumatoid; Rheumatic Diseases; Connective Tissue Diseases; Autoimmune Diseases; Immune System Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- tolerogenic dendritic cells (Experimental): Each dose of autologous monocyte-derived dendritic cells generated in the presence of IFN-α/GM-CSF and tolerized with Dexamethasone (1x106, 3x106, 5x106, 8x106 and 10x106 cells in 2.0 mL sodium chloride 0.9% solution) will be administered in RA patients through intra-articular injection (into the knee joint).
  Interventions: Biological: tolerogenic dendritic cells

INTERVENTIONS:
Biological: tolerogenic dendritic cells — dose-escalation

SUMMARY:
Tolerogenic dendritic cell (tDC)-based clinical trials for the treatment of autoimmune diseases are now a reality. Clinical trials are currently exploring the effectiveness of tDC to treat of type 1 diabetes mellitus, rheumatoid arthritis, multiple sclerosis and Crohn's disease. The general objective of this study is to evaluate the safety and tolerability of a single intra-articular injection (into the knee joint) of autologous monocyte-derived dendritic cells generated in the presence of interferon-alpha (IFN-α)/granulocyte-macrophage colony-stimulating factor (GM-CSF) and tolerized with Dexamethasone in rheumatoid arthritis (RA) patients.

DETAILED DESCRIPTION:
A phase I dose-escalating clinical trial will be conducted to determine the safety and tolerability of a single intra-articular injection (into the knee joint) of autologous tolerogenic dendritic cells, and to enable selection of a suitable dose regimen for phase II trial. The primary objective of the phase I study will be to determine whether tDC-based therapy is safe and well tolerated and to establish the dose-response with disease activity measured over 6 months. Patients will serve as their own controls (pre- and post-treatment). Five doses of tDCs will be tested. The Study will start with intra-articular injection (into the knee joint) of 1x106 cells. Depending on safety/tolerability outcomes, the dose will gradually increase to 3x106, 5x106, 8x106 and 10x106 cells. The safety will be determined by the evaluation of the number of participants with adverse events (AEs) and severe adverse events (SAEs) following the intra-articular administration of tDC (within 6 months of injection). Systemic RA disease activity will be measured using DAS28 (Disease Activity Score using 28 joints) and the Health Assessment Questionnaire (HAQ), a standard instruments used in RA. Patients will be monitored at baseline and at 3, 7 days and 1, 3, 6 months post treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 75 Years
* Patients with moderate to severe active RA (DAS28 >=3.2)
* At least 6 month's disease duration
* Synovitis of large joints (knee, elbow)
* Morning stiffness in the target joint ≥ 30 minutes
* Stable dose of disease-modifying anti-rheumatic drugs (DMARD) for ≥16 weeks
* Patients must be able to tolerate all study procedures
* Patients must be willing to voluntarily give written Informed Consent to participate in the study before any procedures are performed
* Patients must be willing to be available for all baseline, treatment and follow-up examinations required by protocol

Exclusion Criteria:

* Injection of target joint with glucocorticoids within 6 weeks of baseline
* Known hypersensitivity to gentamicin or local anaesthetics
* Dementia, psychiatric disorders
* Renal dysfunctions
* Hemodynamic or respiratory instability
* HIV or uncontrolled bacterial, fungal, or viral infections
* Pregnancy
* Malignancy
* Participation in other clinical trials

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Number of Participants experiencing AEs and SAEs following the intra-articular administration of tDCs. | within 6 months of injection
  Occurrence and severity of adverse events following the intra-articular administration of tDCs will be evaluated within 6 months of injection.

SECONDARY OUTCOMES:
Number of Participants Who Rated the Study and its Components as Partly or Completely Acceptable. | At final study visit, 6 months post treatment
  Participants will assess acceptability of study specific procedures via an "acceptability questionnaire" administered at the last study visit.
Change from Baseline in DAS28 Score. | Baseline, 1, 3 and 6 months post treatment
  DAS28 calculated from the swollen joint count (SJC) and tender joint count (PJC) using the 28 joints count, the erythrocyte sedimentation rate (ESR) (millimeters per hour) and Patient Global Assessment of disease activity (participant-rated arthritis activity assessment) with transformed scores ranging 0 to 10; higher scores indicated greater affectation due to disease activity). A clinically meaningful improvement in DAS28 was defined as an improvement of 1.2 units.
Change from Baseline in the Health Assessment Questionnaire (HAQ) | Baseline, 1, 3 and 6 months post treatment
  Functional status (disability) of participants will be assessed using the Health Assessment Questionnaire (HAQ), a standard instrument used in RA.

CONTACTS AND LOCATIONS:
Overall Officials: Elena R Chernykh, MD, PhD, Study Chair — Institute of Fundamental and Clinical Immunology; Alexander A Ostanin, MD, PhD, Principal Investigator — Institute of Fundamental and Clinical Immunology
Locations (1):
- Institute of Fundamental and Clinical Immunology, Novosibirsk, Russia

IPD SHARING:
Plan to Share IPD: Undecided